CLINICAL TRIAL: NCT00273234
Title: Clinical Evaluation of the Safety and Effectiveness of Topical Autologous Platelet Gel (APG) for the Treatment of Lower Extremity Chronic Venous Insufficiency Ulcers. A Multicenter, Randomized, Controlled Clinical Trial
Brief Title: Clinical Effectiveness of Topical Autologous Platelet Gel for the Treatment of Venous Ulcers
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Lack of financial support. Study criteria severly limited enrollment.
Sponsor: National Healing Corporation (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NHC-2006-01
Record Dates: First submitted 2006-01-04; First posted 2006-01-09 (Estimated); Last update posted 2007-03-06 (Estimated); Status verified 2007-03

CONDITIONS: Venous Ulcer
Keywords: Venous; Ulcer; autologous; platelet; healing
MeSH Terms: conditions — Varicose Ulcer; Ulcer

INTERVENTIONS:
Procedure: Autologous Platelet Gel (APG)

SUMMARY:
The purpose of this study is to compare the effectiveness of standard venous ulcer care to standard venous ulcer care plus a cell based product made from the patients own blood. This product, Autologous Platelet Concentrate (APC), is a concentrate of cells in the bloodstream called platelets.

DETAILED DESCRIPTION:
The purpose of this Pilot clinical study is to make a preliminary clinical and procedural assessment of the treatment of chronic venous stasis ulcers with Autologous Platelet Gel. The information and knowledge gained in the Pilot Study will be used to refine the Investigational Plan under which a Pivotal Clinical Study will be conducted. One of the advantages of conducting a pilot study is that it might give advance warning about where the main research project could fail, where research protocols may not or cannot be followed, or whether proposed methods or instruments are inappropriate or too complicated to achieve the expected clinical outcomes. The Pilot Study will provide preliminary data with which to:

* Assess the feasibility of a (full-scale) study/survey
* Refine the clinical protocol procedures
* Assess the likely success of proposed recruitment approaches
* Identifying logistical problems which might occur using proposed methods
* Estimating variability in outcomes to help determine sample size
* Determine what resources (finance, staff) are needed for a planned study
* Assess the proposed data collection and analysis techniques to uncover potential problems
* Confirm the study objectives are feasible
* Train researcher in the elements of the research process and protocol
* Assess the magnitude of the difference in the effectiveness of the investigational treatment vs control treatment

The pilot study will provide supporting clinical data for an IDE application to FDA for approval to conduct a Pivotal Study of the safety and effectiveness of APG for the treatment of chronic venous stasis ulcers. The study will evaluate the hypothesis that treatment of a chronic venous ulcer with APG prepared from Autologous Platelet Concentrate (APC+) (and the associated autologous growth factors) and Topical Thrombin (TT) has the potential to accelerate the re-epithelialization process. Harvest Technologies will submit a marketing application to FDA to expand the labeling of the SmartPReP2® Platelet Concentrate System, including its accessory kits, with the specific indication to produce APC for the purpose of promoting healing of chronic venous ulcers of the lower extremity.

60 to 100 study subjects will be enrolled from six investigational sites in this single-phase clinical trial.

The SmartPReP®2 Platelet Concentrate System is a dedicated microprocessor-controlled centrifuge. The SmartPReP®2 centrifuge and its accessory, the APC+ Process Kit, are currently available and used to produce Autologous Platelet Concentrate. The Harvest SmartJet Dual Applicator Kit is legally marketed to apply autologous blood products (K000456, K011032, and K020252). Topical Thrombin (TT), (bovine origin), USP is an approved pharmaceutical (NDC 52604-7102-1) marketed by Jones Pharma, Inc. (Thrombin-JMI®) that is not supplied by Harvest and must be obtained by the practitioner.

This study will compare standard of care medical therapy with and without APC+ and TT. Therefore, the study ulcers of the Investigational Group will receive treatment with APC+ and TT as an adjunctive treatment modality in addition to standard therapy.

ELIGIBILITY:
Inclusion Criteria:

* Presence of venous insufficiency lower extremity (below knee) ulcer

  * 4 weeks
* Area of ulcer is 1 cm2 - 20 cm2
* Subject is receiving standard wound care
* ABI ≥ 0.8 or, if diabetic, TBI ≥ 0.8 on the study limb.
* Subject has adequate venous access for phlebotomy.
* Subject has access to reliable outpatient dressing care (self, family member, nursing staff, etc.)
* Hematocrit is > 30%
* Platelet Count is > 100,000
* INR < 1.3
* Subject has no known coagulopathies
* Serum Albumin > 2.5
* If diabetic, HgbA1C < 10%
* Venous reflux < 20 seconds by ultrasonography

Exclusion Criteria:

* Presence of arterial insufficiency (ABI or if diabetic TBI <0.8)
* Subject has received biological therapy within 30 days of enrollment
* Subject is receiving radiation therapy near the ulcer
* Active infection of the study wound, or osteomyelitis, or cellulitis has been diagnosed. The patient may be enrolled only after the infection has been controlled, including:
* Debridement if necessary
* Patient has received at least 2 weeks of appropriate antibiotics
* Allergy to bovine thrombin
* Alcohol or drug abuse within 6 months of enrollment
* Subject has been diagnosed with AIDS, HIV, or Hepatitis
* Subject is taking immunosuppressive therapy
* Subject is taking pentoxyfilline (Trental®)
* Steroid use within 7 days of enrollment
* Presence of a non-study ulcer within 2.0cm of the study ulcer
* Angioplasty by bypass or endovascular therapy within 4 weeks of enrollment
* Suspected sleep apnea
* Active Cancer
* BMI > 40 kg/m2
* Severe Rheumatoid Arthritis
* Collagen vascular disease
* Female who is pregnant or lactating or not using a reliable birth control method if of child-bearing age
* Wound bed with exposed bone, tendon, or fascia
* Renal insufficiency defined as Creatinine > 3 mg/dL
* Hepatic insufficiency defined as total Bilirubin > 2 mg/dL
* Enrollment, within the past 3 months, in any study related to wound healing
* Closure of study wound ≥ 40% within 2 screening visits of enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70
Dates: Start 2006-01; Study Completion 2006-11

PRIMARY OUTCOMES:
Complete Healing

SECONDARY OUTCOMES:
Percent Healing per unit of time (speed)
Pain reduction

CONTACTS AND LOCATIONS:
Overall Officials: Bob Bartlett, MD, Principal Investigator — National Healing Corporation; Steve Martin, PhD Candidate, Health Science, Principal Investigator — Touro University International
Locations (6):
- United States (6):
  - Palms of Pasadena Wound Healing Center, St. Petersburg, Florida
  - Parrish Wound Healing Clinic, Titusville, Florida
  - Anna Jacques Hospital Wound Healing Center, Newburyport, Massachusetts
  - Johnston Therapeutic Wound Clinic, Smithfield, North Carolina
  - Ohio State University East Wound Healing Center, Columbus, Ohio
  - East Texas Medical Center Wound Healing Center, Tyler, Texas